CLINICAL TRIAL: NCT00841607
Title: Reconstruction Following Pancreaticoduodenectomy: A Randomized Clinical Trial of Pancreaticojejunostomy vs Pancreaticogastomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tom Baker Cancer Centre (Other)
Collaborators: MSI Foundation (Unknown); University of Calgary (Other); Canadian Association of General Surgeons (Other)
Responsible Party: Principal Investigator, Elijah Dixon, Professor of Surgery, Oncology and Community Health Sciences, Tom Baker Cancer Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18982
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Pancreas Cancer; Periampullary Cancer
Keywords: whipple; pancreas; reconstruction; leak; fistula
MeSH Terms: conditions — Pancreatic Neoplasms; Fistula

ARMS (2):
- Pancreaticojejunostomy (Experimental): Pancreaticojejunostomy reconstruction used following Whipple surgery.
  Interventions: Procedure: pancreaticojejunostomy vs pancreaticogastrostomy
- Pancreaticogastomy (Active Comparator): Pancreaticogastomy reconstruction used following Whipple surgery.
  Interventions: Procedure: pancreaticojejunostomy vs pancreaticogastrostomy

INTERVENTIONS:
Procedure: pancreaticojejunostomy vs pancreaticogastrostomy

SUMMARY:
Pancreaticoduodenectomy (PD or Whipple procedure) involves the removal of the head of the pancreas and is the primary modality for treatment of peri-ampullary cancers (arising from the common bile duct, Ampulla of Vater, duodenum, neuroendocrine cells of the pancreas, and most commonly the exocrine pancreas). In Canada, cancer of the pancreas is the 11th cancer in terms of new cases/year, and the 5th leading cause of cancer related deaths/year. Following PD the remaining pancreas is re-connected to a portion of the gastrointestinal tract; the pancreas is very soft and difficult to sew and connect safely. The primary cause of complications following PD is related to leak occurring at this connection. Of patients that develop a leak, over half need a second operation, and up to 40% will die. The two main organs that the pancreas may be re-connected to are the jejunum or the stomach. The investigators will compare the rates of pancreatic leakage in two groups of patients randomized to reconnection to either the jejunum or stomach following PD. The goal of this study is to determine which of these methods is safer. The results may change practice patterns across North America and the world. It may in the future prevent many cases of avoidable leakage and the resulting morbidity of this including death. This will therefore reduce the morbidity and mortality of this group of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Suspected pancreatic or periampullary neoplasm that appears to be resectable based on preoperative imaging (CT scan and/or MRI) and are deemed medically fit to undergo PD.

Exclusion Criteria:

* Patients less than 18 years of age will be excluded.
* As well, patients with distant metastasis, local unresectability, and/or gastric involvement will be excluded.

Other exclusion criteria include:

* female subjects who are pregnant or nursing
* current use of an investigational drug
* currently receiving chemotherapy or radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2006-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
pancreatic leak/fistula | Up to POD 10
  Either a radiologically proved anastomotic leak or the continued drainage (via drain, enterocutaneous fistula, or wound) of amylase (or lipase) rich fluid on or after postoperative day 10. This is a clinically relevant definition which has been used in many other reports.

SECONDARY OUTCOMES:
overall morbidity | Up to POD 30
  We will use the definition and classification of complications resulting from surgery as put forth by Clavien et al which has been widely adopted in the surgical literature.

CONTACTS AND LOCATIONS:
Overall Officials: elijah dixon, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Background] McKay A, Mackenzie S, Sutherland FR, Bathe OF, Doig C, Dort J, Vollmer CM Jr, Dixon E. Meta-analysis of pancreaticojejunostomy versus pancreaticogastrostomy reconstruction after pancreaticoduodenectomy. Br J Surg. 2006 Aug;93(8):929-36. doi: 10.1002/bjs.5407. PMID 16845693
- [Derived] Grendar J, Ouellet JF, Sutherland FR, Bathe OF, Ball CG, Dixon E. In search of the best reconstructive technique after pancreaticoduodenectomy: pancreaticojejunostomy versus pancreaticogastrostomy. Can J Surg. 2015 Jun;58(3):154-9. doi: 10.1503/cjs.010014. PMID 25799130